CLINICAL TRIAL: NCT04336748
Title: Low-dose Hydroxychloroquine for Primary Prophylaxis Against SARS-CoV-2 in Health-care Workers - a Randomized, Double-blind, Controlled Trial
Brief Title: HCQ for Primary Prophylaxis Against COVID19 in Health-care Workers
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not feasible
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Matthias Vossen, Priv. Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HCQ prophylaxis for COVID19
Record Dates: First submitted 2020-04-04; First posted 2020-04-07 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Sars-CoV2; Infection Viral; Healthcare Worker; Prophylaxis
MeSH Terms: conditions — Virus Diseases | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (Active Comparator): 200mg once daily
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — low dose (200mg) Hydroxychloroquine once daily for 4 weeks
  Arms: Hydroxychloroquine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Background:

Aim: To demonstrate the efficacy of low-dose hydroxychloroquine as primary prevention in healthcare workers Design, participants and interventions: Prospective, randomized, parallel group, double-blinded, placebo controlled, study.

including 440 participants who will be randomised to 2 treatment arms: hydroxychloroquine or placebo.

Outcome variables: symptomatic or asymptomatic SARS-CoV-2 infection confirmed by PCR, viral load during SARS-CoV-2 infection, seroconversion during the study period, incidence of any acute respiratory infection, days of sick leave.

Statistical considerations: No trials have been published investigating the efficacy of HCQ as primary prophylaxis of SARS-CoV-2 infection in health care workers. Thus, sample size calculations in the proposed trial are based on the investigators' best estimates for several parameters.

In accordance to the effect of oseltamivir against symptomatic influenza, we assumed an approximate effectiveness of approximately 60% (HR of 0.4) (https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6464969/) as realistic. As a prophylactic intervention with HCQ, which may have side effects and for which supply shortage can be expected, was judged justifiable only if its effectiveness is high, we based our sample size consideration on a HR of 0.3. To estimate the probability of an event in both the experimental and the control group, very little data is available. In a Dutch point-prevalence study 0-10% of health-care workers were infected depending on the healthcare institution, depending on the hospital. This point-prevalence study was performed between 6 and 9 March, when the reported number of cases in the Netherlands was 33 and 77, respectively, according to the RIVM (https://www.rivm.nl/nieuws/resultaat-steekproef-4-ziekenhuismedewerkers-heeft-coronavirus). Additionally, in an a report published in the Lancet, 20% of responding healthcare workers in Italy were found to be infected with SARS-CoV2 within less than one month (https://www.thelancet.com/journals/lancet/article/PIIS0140-6736(20)30627-9/fulltext). Several media reports indicate that this proportion is similar across various healthcare institutions and countries (https://www.nytimes.com/2020/03/24/world/europe/coronavirus-europe-covid-19.html) and (https://www.aljazeera.com/news/2020/03/spain-tightens-restrictions-week-lockdown-begins-200330191539568.html).

As the proposed study will be performed in a high-risk setting, we assumed an event (i.e. PCR positivity) probability of 10% in the control group and 3% in the experimental arm after the maximum study period. In summary, a sample size of 210 participants per arm is necessary to detect a HR of 0.3 with a power of 80.3% with an alpha-error of 0.05. To account for drop-outs and asymptomatic, undetected infection at inclusion or past infection with existing immunity, an additional 10 participants will randomized per treatment arm. The overall study population is therefore 440 participants.

Statistical analysis will be based on two populations: A Modified Intention to Treat population excluding those who withdrew consent after randomization and those with a positive serology at baseline. And a per protocol population including all randomized subjects who completed at least 3 out of 4 follow-up visits and took at least 80% of all doses of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Health-care worker with frequent contact with confirmed COVID-19 patients
* No active or past infection with SARS-CoV-2
* 18 years of age or older
* No allergy or contraindication to hydroxychloroquine
* written informed consent

Exclusion Criteria:

* Age of less than 18 years
* Pregnancy or lactation
* unwillingness to use effective contraception during the participation in the trial
* Use of concomitant medication that prolongs the QT interval
* Allergy or contraindication to hydroxychloroquine
* Retinopathy or maculopathy
* Neuromuscular diseases (i.e Myasthenia gravis, Parkinson's disease)
* G6PD Deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Symptomatic or asymptomatic SARS-CoV-2 infection confirmed by PCR | 4 weeks

SECONDARY OUTCOMES:
Viral load during SARS-CoV-2 infection | 4 weeks
Seroconversion during the study period | 4 weeks
Incidence of any acute respiratory infection | 4 weeks
Days of sick leave | 4 weeks